CLINICAL TRIAL: NCT05775237
Title: An Open-Label, Three-Arm, Parallel, Investigator-Initiated Trial of Three Different Gummies (Curcumin Gummies, Vitamin C Gummies, and Vitamin B Complex Gummies) in Healthy Children
Brief Title: An Investigator-initiated Trial to Assess the Effectiveness of Three Different Gummies (Curcumin Gummies, Vitamin C Gummies, and Vitamin B Complex Gummies) in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Responsible Party: Principal Investigator, Dr Chitra Prajapati, Principal Investigator, NeighbourCare Clinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NB230001-NCP
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Healthy Children
MeSH Terms: interventions — Curcumin; Ascorbic Acid; Geritol

STUDY DESIGN:
Intervention Model Description: An Open-Label, Three-Arm, Parallel, Investigator-Initiated Trial of clinical study
Masking Description: This Study is Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Curcumin Gummies (Experimental): Curcumin Gummies contain energy, dietary fiber, sugar, total carbohydrate, protein, fat, and curcumin.
  Interventions: Dietary Supplement: Curcumin Gummies
- Vitamin C Gummies (Experimental): Vitamin C Gummies contain Vitamin C and Zinc
  Interventions: Dietary Supplement: Vitamin C Gummies
- Multivitamin Gummies (Experimental): Multivitamin Gummies contain energy, dietary fiber, sugar, total carbohydrate, protein, fat, sodium, Vitamin C, Vitamin E, pantothenic acid, Zinc, iodine, Vitamin A, Magnesium, Folate, Vitamin D, Vitamin 12
  Interventions: Dietary Supplement: Multivitamin Gummies

INTERVENTIONS:
Dietary Supplement: Curcumin Gummies — Chew gummies thoroughly and completely before swallowing.
  Other Names: curcumin
  Arms: Curcumin Gummies
Dietary Supplement: Vitamin C Gummies — Chew gummies thoroughly and completely before swallowing.
  Other Names: Vitamin C
  Arms: Vitamin C Gummies
Dietary Supplement: Multivitamin Gummies — Chew gummies thoroughly and completely before swallowing.
  Other Names: Multivitamin
  Arms: Multivitamin Gummies

SUMMARY:
An Open-Label, Three-Arm, Parallel, Investigator-Initiated Trial of Three Different Gummies (Curcumin Gummies, Vitamin C Gummies, and Vitamin B Complex Gummies) in Healthy Children.

A sufficient number (maximum of 48, (16 children/arm)) of children subjects will be recruited to ensure a total of 45 subjects (15 children /arm) complete the study.

DETAILED DESCRIPTION:
Qualifying siblings within the same household are permitted in the study. The potential subjects will be screened as per the inclusion and exclusion criteria only after obtaining written parental informed consent and from the subjects and subjects' legal parent/legal guardian.

The subject's parents will be instructed to visit the facility as per the below visits:

* Visit 01 (Day 01): Screening, Enrolment Visit
* Visit 02 (Day 30): Evaluations, End of Study Visit Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be called on the telephone by the recruiting department prior to the enrolment visit.

Assessment of safety, efficacy and organoleptic properties will be done on Day 01 as a baseline before test product usage to Day 30 after test product usage.

Reduction in frequency of getting the sickness. Consumer feedback-subjective questionnaires - Health Questionnaire Product Perception Questionnaire - Organoleptic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 02 to 12 years old (both inclusive) at the time of parental consent.
2. Overall good health of the child subject is determined by medical examination and history evaluated by the Investigator.
3. Subject's mother/legal guardian, preferably willing to give a voluntary written informed consent i.e. parental informed consent form and agree to complete study activities and come for regular follow-up with a subject.
4. The subject's mother/legal guardian for their child is preferably willing to abide by and comply with the study protocol.
5. The subject should not participate in any other clinical study during participation in the current study
6. Subject are agreed to maintain current level of activity through the study.

Exclusion Criteria:

1. Subjects with known history of allergies or specific allergic reactions upon using curcumin, vitamins, zinc, pantothenic acid.
2. Subjects who are currently enrolled in an active investigational study or have participated in an investigational study within 30 days prior to enrolment.
3. Subjects, who in the opinion of the Investigator or the Expert physician are not eligible for enrolment in the study.
4. Subject who are unwilling to provide consent.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety | Day 01 before test product usage to 30 Day after Test product usage
  To evaluate the Safety of Test Product by using subject perception questionnaires regarding Health
Assessment of Efficacy | Day 01 before test product usage to 30 Day after Test product usage
  To evaluate the Efficacy of Test Product by using subject perception questionnaires regarding Health
Assessment of Organoleptic properties | 30 Day after usage of Test product
  To evaluate the Organoleptic properties of Test Product by using subject perception questionnaires regarding Test Product

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Chitra Prajapati, MBBS, Principal Investigator — Principal Investigator
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No